CLINICAL TRIAL: NCT02854215
Title: Cost Utility of Radical Surgery in Ovarian Cancer
Acronym: CURSOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15GENF03
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian cancer (Other): Patient undergoing primary surgery for a newly diagnosed ovarian, tubal or peritoneal malignancies; Stage IIIc or IVa with extrapelvic carcinomatosis according to the International Federation of Gynecology and Obstetrics classification 2014
  Interventions: Other: Collection of additional data with questionnaires

INTERVENTIONS:
Other: Collection of additional data with questionnaires — * questionnaires for quality of life measurements: QLQC30; QLQ-OV28
  * questionnaires for medico-economic purposes: ADL (activities of daily living); IADL (instrumental activities of daily living); EQ-5D3L; absenteeism questionnaire.
  These questionnaires will be completed during the study time (5 or 6 times during the treatment, next every 4 months during the first two years and then every 6 months during the third year of follow-up).

SUMMARY:
The purpose of this study is to investigate the medico-economic impact of adherence to INCa (National Cancer Institute) guidelines in ovarian cancer surgery by assessment of outcome in cost per Quality Adjusted Life Years (QALY).

DETAILED DESCRIPTION:
This is a prospective, multicenter, comparative and non-randomized study designed to investigate the medico-economic impact of adherence to INCa guidelines in ovarian cancer surgery by assessment of outcome in cost per Quality Adjusted Life Years (QALY).

A cost-utility study will be performed. It will primarily aim to assess the Incremental Cost-Utility Ratio (ICUR) at 3 years of the two treatment strategies of ovarian cancer surgery: adherence to INCa quality indicators versus non-adherence to INCa quality indicators.

Consecutive patients with stage IIIC and IV ovarian, tubal, and primary peritoneal malignancies will be recruited in different health care institutions, including comprehensive cancer centers, university hospitals and private hospitals.

Evaluation of adherence to quality indicators will be assessed retrospectively (once patients have completed the treatment) by two independent experts.

200 patients will be included over a period of 2 years and will be followed for a 3 years period after treatment (every 4 months the first two years and then every 6 months).

ELIGIBILITY:
Inclusion Criteria:

* 1. Woman with age ≥ 18 years.
* 2. Newly diagnosed ovarian, tubal or peritoneal malignancies.
* 3. Epithelial histology.
* 4. Stage IIIC or IVA with extrapelvic carcinomatosis according to FIGO classification 2014.
* 5. Patients undergoing primary surgery or neoadjuvant chemotherapy.
* 6. Performance Status ≤ 2.
* 7. Patient affiliated to a Social Health Insurance in France.
* 8. Patient information and informed consent form signed prior to any study specific procedures.

Exclusion Criteria:

* 1. Benign or borderline tumors.
* 2. Patients with extra-abdominal disease, except for pleural effusion with positive cytology.
* 3. Other malignancy diagnosed in the previous 5 years except skin cancer (other than melanoma).
* 4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
* 5. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Cost-utility study | 5 years and 6 months
  The primary endpoint is defined as cost per Quality-Adjusted Life Year (QALY) at 3 years. Patient utilities will be obtained from the EuroQoL 5D-3L questionnaire.

SECONDARY OUTCOMES:
Rate of institutions adherent to INCa quality indicators | 2 years and 6 months
  The rate of institutions adherent to INCa quality indicators corresponds to the number of institutions adherent to INCa quality indicators among the total number of institutions.
Rate of patients "adherent" to INCa quality indicators | 2 years and 6 months
  The rate of patients "adherent" to INCa quality indicators corresponds to the number of patients adherent to INCa quality indicators among the total number of patients.
Quality of life | 5 years and 6 months
  The quality of life will be evaluated according to the QLQ-C30, QLQ-0V28 and the EQ-5D-3L questionnaires
Budgetary impact on the health insurance budget of these INCa quality indicators on the care management of ovarian cancer patients | 5 years and 6 months
  Budgetary impact on the health insurance budget of these INCa quality indicators on the care management of ovarian cancer patients using costs data collected from the French insurance databases, Medical Information Departments of each participating centers and from patients' questionnaires (treatment costs, other induced costs and avoided costs).
Progression Free Survival | 5 years and 6 months
  Progression Free Survival is defined as the time from inclusion until progression or death from any cause
Overall Survival | 5 years and 6 months
  Overall Survival is defined as the time from inclusion until death from any cause or last follow-up news (censored data).
Morbidity | 5 years and 6 months
  Morbidity will be assessed through recording of adverse events using NCI-CTCAE toxicity classification and vital signs measurement.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut Bergonie, Bordeaux
  - Chu Clermont Ferrand, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Paoli Calmettes, Marseille
  - Institut Regional Du Cancer Montpellier, Montpellier
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud 1, Pierre-Bénite
  - Centre Hospitalier Lyon Sud 2, Pierre-Bénite
  - Institut Claudius Regaud, Toulouse
  - Hopital Nord-Ouest - Villefranche Sur Saone, Villefranche-sur-Saône

REFERENCES:
- [Derived] Filleron T, Lusque A, Dalenc F, Ferron G, Roche H, Martinez A, Jouve E. Alternative methodological approach to randomized trial for surgical procedures routinely used. Contemp Clin Trials. 2018 May;68:109-115. doi: 10.1016/j.cct.2018.03.016. Epub 2018 Mar 30. PMID 29608972